CLINICAL TRIAL: NCT04309760
Title: Developmental Correlates and Hormone Therapy Effects in Gender Dysphoria
Acronym: DCHGD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the patients are now followed in another hospital. The study is discontinued
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A01997-50
Record Dates: First submitted 2020-02-18; First posted 2020-03-16 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Gender Dysphoria
Keywords: gender dysphoria; neuroimaging; hormone-surgical reassignment
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Intervention Model Description: Comparison between Mtf and control subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gender dysphoria subjects (Active Comparator): Patients with MtF gender dysphoria (biological men who are transitioning to the female gender) attending the forensic psychiatric consultation for a request for hormone-surgical reassignment. Subjects will receive initial clinical assessment and MRI before and 6 months after initiation of hormone therapy
  Interventions: Other: MRI
- control subjects (Other): Control group inclusions, of open-label patients without gender dysphoria.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Subjects will receive structural and functional (resting state) MRI

SUMMARY:
The aim of the research is to study longitudinally the effects of reassignment hormonotherapy on the connectome of MtF (biological men who are transitioning to the female gender) dysphoric subjects after 6 months of hormone therapy. The subjects will be compared to a control group of healthy subjects taking into account sexual orientation

DETAILED DESCRIPTION:
The pathophysiology of gender dysphoria is still poorly understood, but a number of clues point to an origin derived from biological and environmental factors, particularly studies of twins, birth order, and family groups. Several explanatory models have been put forward. In particular, the differentiation of genitals taking place in the first half of pregnancy while that of the brain in the second makes it possible to imagine a different differentiation between the external phenotype and the cerebral gender. Several developmental features have thus been found in gender dysphoric subjects, including the finger length ratio D2 / D4, lateralization. Some neuroimaging studies have shown brain features in gender dysphoric subjects that seem original compared to control subjects. Nevertheless, the results are scarce, poorly reproduced, and for some, the differences highlighted may be related to phenotypic variability including the non-consideration of sexual orientation. Moreover, some of these studies combine subjects treated or not with hormone therapy which is a bias because it is likely that hormone therapy may have structural and functional effects on brain function. The investigators team deals with dysphoric gender issues as part of a coordinated course of hormone-surgical reassignment. We wish to better characterize the brain effects, at the level of the "connectome" of the reassignment hormone therapy in a population of dysphoric subjects, taking into account signs of pre-natal hormonal impregnation (D2 / D4 ratio), developmental features (onset of dysphoria, lateralization, size), and controlling sexual orientation as a potential confounding factor.

The aim of the research is then to study longitudinally the effects of reassignment hormonotherapy on the connectome of MtF dysphoric subjects after 6 months of hormone therapy. The subjects will be compared to a control group of healthy subjects taking into account sexual orientation.

This is a prospective longitudinal study that includes, in a consecutive manner, open-label patients with MtF gender dysphoria (biological men who are transitioning to the female gender) attending the forensic psychiatric consultation for a request for hormone-surgical reassignment. Subjects will receive initial clinical assessment and MRI before and 6 months after initiation of hormone therapy; the imaging data will be compared to a control group (n = 20).

ELIGIBILITY:
Inclusion Criteria:

* gender dysphoric subjects MtF
* right handed
* androphilic orientation
* without hormone therapy

Control group of male subjects:

* right handed
* without any psychiatric or medical history
* androphilic orientation

Exclusion Criteria:

* MRI contraindication
* vulnerable adults
* mental retardation
* psychiatric or neurological disease including autism spectrum disorders, psychotropic medication
* hormonal or genetic condition

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Brain connectome 6 months after the hormone therapy beginning | 6 months after the beginning of the hormone therapy
  Structural and functional MRI before and after 6 months of hormone therapy will be analysed in order to make a comparison before/after

SECONDARY OUTCOMES:
Brain connectome in gender dysphoric and control subjects | baseline
  The MRI images will be analysed in order to construct a brain " connectome " which reflects brain connectivity, using the graph theory. At baseline, these networks will be compared between dysphoric and control subjects.
Gender dysphoria phenotype description | baseline and 6 months after the beginning of the hormone therapy
  The MRI images will be analysed in order to construct a brain " connectome " which reflects brain connectivity, using the graph theory. Correlations will be made at baseline between brain connectome of the dysphoric subjects and testosteronemia, and developmental measures : age at beginning of gender dysphoria, finger lenghth D2/D4 ratio, birth weight, laterality using Edimbourg scale.
Brain connectome variations | 6 months after the beginning of the hormone therapy
  The MRI images will be analysed in order to construct a brain " connectome " which reflects brain connectivity, using the graph theory. Evolutions of the brain connectome of dysphoric subjects will be compared after 6 months of hormone therapy, taking into acount gender dysphoria decrease measured using Utrecht Gender Dysphoria Scale.

IPD SHARING:
Plan to Share IPD: Undecided